CLINICAL TRIAL: NCT02320617
Title: Application of Diffusion Weighted Magnetic Resonance Imaging Versus CT in Evaluation of the Effect of Treating Lung Cancer
Brief Title: Application of Diffusion Weighted MRI Versus CT in Evaluation of the Effect of Treating Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Jian Zhang, deputy director of department of respiratory medicine, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013C2014
Record Dates: First submitted 2014-12-09; First posted 2014-12-19 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Lung Neoplasms
Keywords: Lung Neoplasms; diffusion weighted MRI; ADC value; treatment effect
MeSH Terms: conditions — Lung Neoplasms | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DW-MRI group (Experimental): To evaluate the efficacy of chemoradiotherapy in lung cancer patients by DW-MRI when compared with conventional imaging modalities(CT, ultrasound et al.)
  Interventions: Procedure: Diffusion Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Diffusion Magnetic Resonance Imaging — Diffusion weighted imaging (DWI) is a form of magnetic resonance imaging based upon measuring the random Brownian motion of water molecules within a voxel of tissue. The relationship between histology and diffusion is complex, however generally densely cellular tissues or those with cellular swelling exhibit lower diffusion coefficients, and thus diffusion is particularly useful in tumour characterisation
  Other Names: DW-MRI

SUMMARY:
The purpose of this study is to investigate the diagnostic accuracy of ADC value of diffusion weighted MRI in comparison of conventional treatment assessment criteria in evaluation of chemotherapy. Moreover, the investigators aim to clarify the correlation of ADC value with histologic type and grade of lung cancer and survival of patients.

DETAILED DESCRIPTION:
In recent years, lung cancer is an aggressive and heterogeneous disease, Advances in surgical and chemotherapeutic approaches have been made, but the long-term survival rate remains low. Although effective mass screening of high-risk groups could potentially be of benefit, randomized trials of screening with the use of chest radiography with or without cytological analysis of sputum specimens have shown no reduction in lung-cancer mortality. Currently, Response Evaluation Criteria in Solid Tumors (RECIST) by CT is the most commonly used to evaluate chemotherapy of lung cancer patient, but patients have to be exposed to radiation. For this reason, the investigators aim to assess the diagnostic accuracy of apparent diffusion coefficient (ADC) value, a specific parameter of radiation-free diffusion weighted MRI, in comparison of RECIST, and its correlation with histologic type and grade of lung cancer as well. Furthermore, the investigators investigate its correlation with Progression Free Survival (PFS) and Overall Survival (OS) in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75
2. Patients have confirmed lung cancer by histopathological methods (fiber, bronchoscopy, lung biopsy, open chest biopsy, pleural effusion exfoliated cells, sputum exfoliated cells)
3. After clinical assessment, patients who need chemotherapy (tumor stage III or IV of lung cancer or others who are reluctant to receive pneumonectomy);
4. Patients have no previous history of chemotherapy
5. Patients with at least one clearly measurable lung lesion (lesion size larger than 10mm, by spiral CT, according to RECIST)
6. Health status scoring between 0-2 by Eastern Cooperative Oncology Group(ECOG) method
7. Patients voluntarily to join this study and signed informed consents.

Exclusion Criteria:

1. Any body metal implants (pacemaker implantation, nerve stimulator, vascular stent, aneurysm clip, eye foreign body, the inner metal prosthesis) or artificial heart valves
2. Patients with claustrophobia to MRI or CT examination
3. Patients who are reluctant to comply with follow-up and subsequent examination
4. The other condition that do not meet the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-11 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ADC value | 4,8,12 weeks post initial chemotherapy
  Change from baseline in ADC value in 4,8,12 weeks(every two cycles of chemotherapy) post initial treatment when compared with RECIST (based on the CT examination), thus it can be estimated that the accuracy of ADC value in evaluating chemotherapy.

SECONDARY OUTCOMES:
ADC value | 1 day before initial chemotherapy
  The correlation of ADC value in 1 day before initial chemotherapy with histologic type and grade of lung cancer

OTHER OUTCOMES:
Change from baseline in ADC value | At the date of first documented progression, assessed up to 12 months
  Change from baseline in ADC value will be documented at date of first documented progression, assessed up to 12 months post initial chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jian, professor, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Honda O, Tsubamoto M, Inoue A, Johkoh T, Tomiyama N, Hamada S, Mihara N, Sumikawa H, Natsag J, Nakamura H. Pulmonary cavitary nodules on computed tomography: differentiation of malignancy and benignancy. J Comput Assist Tomogr. 2007 Nov-Dec;31(6):943-9. doi: 10.1097/RCT.0b013e3180415e20. PMID 18043361
- [Result] Zhang J, Cui LB, Tang X, Ren XL, Shi JR, Yang HN, Zhang Y, Li ZK, Wu CG, Jian W, Zhao F, Ti XY, Yin H. DW MRI at 3.0 T versus FDG PET/CT for detection of malignant pulmonary tumors. Int J Cancer. 2014 Feb 1;134(3):606-11. doi: 10.1002/ijc.28394. Epub 2013 Sep 16. PMID 23893610